CLINICAL TRIAL: NCT05046483
Title: Metabolic Phenotyping and Follow-Up of Patients With and Without Diabetes Mellitus After New Onset of ST-Segment Elevation Myocardial Infarction (STEMI) (DISTEMI Study)
Brief Title: Metabolic Phenotyping and Follow-Up of Patients With and Without Diabetes After New Onset of STEMI
Acronym: DISTEMI
Status: Recruiting | Type: Observational
Sponsor: German Diabetes Center (Other)
Responsible Party: Sponsor
Other Study IDs: DISTEMI-Study-01
Record Dates: First submitted 2021-09-07; First posted 2021-09-16 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: ST-segment Elevation Myocardial Infarction (STEMI); Diabetes Mellitus; Insulin Resistance; Non-Alcoholic Fatty Liver Disease
Keywords: ST-segment elevation myocardial infarction; STEMI; Cardiovascular diseases; CVD; Diabetes mellitus; Normal glucose tolerance; Non-alcoholic fatty liver disease; NAFLD; Liver fibrosis
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Diabetes Mellitus; Insulin Resistance; Non-alcoholic Fatty Liver Disease; Cardiovascular Diseases; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole-blood, peripheral blood mononuclear cells, serum, plasma, urine, stool
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort with type 1 diabetes (T1D) and type 2 diabetes (T2D): Prospectively followed cohort of people with new onset of ST-segment elevation myocardial infarction and diabetes mellitus (type 1 or type 2) according to the American Diabetes Association (ADA) and German Diabetes Society (DDG) criteria (HbA1c ≥6.5% or pathological oral glucose tolerance test (OGTT)), aged 18-80 years at inclusion into the study
- Cohort of normal glucose tolerant people (NGT): Prospectively followed cohort of healthy people with new onset of ST-elevation myocardial infarction and normal glucose tolerance status (HbA1c <5.7% and normal OGTT), aged 18-80 years at inclusion into the study
- Cohort of people with impaired glucose metabolism (IGM): Prospectively followed cohort of people with new onset of ST-elevation myocardial infarction and impaired glucose metabolism, usually called prediabetes including impaired fasting glucose (IFG) and/or impaired glucose tolerance (IGT) and/or HbA1c 5.7-6.4%, aged 18-80 years at inclusion into the study

SUMMARY:
The aim of the prospective observational DISTEMI-Study in people with and without Diabetes mellitus (DI) after new onset of ST-Segment Elevation Myocardial Infarction (STEMI) aged 18-80 years at inclusion into the study is to characterize in detail the clinical, metabolical, immunological and vascular phenotype, investigate the interplay between myocardial remodelling and the metabolic phenotype, monitor the progression of the disease and compare the phenotype of STEMI people with diabetes mellitus to people with prediabetes and glucose tolerant people.

DETAILED DESCRIPTION:
In detail, the following questions will be answered:

1. Do distinct metabolic phenotypes (with respect to insulin secretion, insulin sensitivity, circulating free fatty acids and ectopic lipid storage, especially in the liver) determine myocardial infarct size and decline of contractile function of the remote myocardium?
2. Which factors modify the progression of the disease (insulin resistance, ectopic lipid storage, subclinical inflammation, abnormal energy metabolism)? People are thoroughly examined at baseline and one year after STEMI.
3. Can we identify risk profiles and their relevance for development of diabetes-associated complications as well as long-term progression of diabetes?
4. Can we improve risk assessment algorithms for targeted therapy in line with Precision Medicine?

ELIGIBILITY:
Inclusion Criteria:

* Condition after new onset of ST-segment elevation myocardial infarction (STEMI)
* Age 18-80 years
* HbA1c <9.0%
* People with diagnosis of diabetes mellitus according to ADA and DDG criteria (i.e. HbA1c ≥6.5% and/or pathological oral glucose tolerance test)
* Healthy people with normal glucose tolerance status according to ADA and DDG criteria (i.e. HbA1c <5.7% and normal OGTT)
* People with impaired glucose metabolism ("prediabetes") according to ADA and DDG criteria (i.e. impaired fasting glucose and/or impaired glucose tolerance and/or HbA1c 5.7-6.4%)
* Consent-able, hemodynamically stable people, without sedation (e.g. opiates) or other interfering medication (e.g. catecholamines)

Exclusion Criteria:

* Diabetes mellitus category 3 A-H (ADA criteria), gestational diabetes
* Current pregnancy
* Infectious diseases, acute infections / fever
* Immunosuppressive therapy
* Severe chronic renal, liver or heart disease (e.g. serum creatinin ≥1.6 mg/dl, peripheral artery occlusive disease stage IV)
* Malignant diseases
* Severe chronic psychiatric illness or addiction
* Participation in an intervention trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Maximum care hospital: Department of Cardiology, Pumonology and Vascular Medicine at University Hospital Düsseldorf (UKD), Heinrich Heine University (HHU), Düsseldorf.
  People with STEMI are recruited by screening at the German Diabetes Center (GDC/DDZ), Institute for Clinical Diabetology, Leibniz Institute for Diabetes Research at HHU Düsseldorf.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-12-30 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Change of cardiac function | One year
  Measurement of left-ventricular ejection fraction by cardiac magnetic resonance (MR) imaging

SECONDARY OUTCOMES:
Change of insulin sensitivity (M-Value) | One year
  Measurement of whole body insulin sensitivity with hyperinsulinemic euglycemic clamp (HEC)
Change of insulin secretion | One year
  Measurement of beta-cell function with oral and intravenous glucose tolerance test
Change of ectopic fat distribution | One year
  Measurement of cardiac and hepatic lipid content by MR spectroscopy (MRS)
Change of liver stiffness | One year
  Measurement of liver stiffness by transient elastography (Fibroscan®) and MR elastography (MRE)
Change of energy metabolism | One year
  Measurement of myocardial and hepatic phosphocreatine(PCr)-to-adenosine triphosphate(ATP) Ratio by MRS
Change of mitochondrial respiratory function | One year
  Measurement of lymphocyte mitochondrial respiration by Oxygraph-O2k
Change of Fatty liver index | One year
  Estimate calculated by laboratory and anthropometric parameters for assessment of liver steatosis
Change of Homeostasis Model Assessment 2 Estimate | One year
  HOMA2-IR is calculated by laboratory and anthropometric parameters for non-invasive assessment of insulin sensitivity under fasted condition
Incidence of further cardiovascular diseases (CVD) and STEMI-related complications, new onset of prediabetes and diabetes mellitus and associated comorbidities | One year
  Determination of the prevalence of cardiovascular diseases and associated complications (i.e. heart failure, recurrent infarction, morbidity, mortality), new onset of prediabetes and diabetes, diabetes-related complications and associated comorbidities

CONTACTS AND LOCATIONS:
Overall Officials: Michael Roden, Prof., MD, Principal Investigator — German Diabetes Center
Locations (1):
- German Diabetes Center, Düsseldorf, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Heilmann G, Trenkamp S, Moser C, Bombrich M, Schon M, Yurchenko I, Strassburger K, Rodriguez MM, Zaharia OP, Burkart V, Wagner R, Roden M. Precise glucose measurement in sodium fluoride-citrate plasma affects estimates of prevalence in diabetes and prediabetes. Clin Chem Lab Med. 2023 Oct 24;62(4):762-769. doi: 10.1515/cclm-2023-0770. Print 2024 Mar 25. PMID 37870928